CLINICAL TRIAL: NCT04797351
Title: Acceptability and Feasibility of a DBT Skills Group Intervention for Bipolar Disorder - a Randomized Pilot Trial
Brief Title: Bi-REAL - DBT Skills Online Group Intervention for Bipolar Disorder
Acronym: BI-REAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Julieta Azevedo (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other); ADEB - Associação de Apoio a Doentes Depressivos e Bipolares (Unknown); Unidade Local de Saúde de Coimbra, EPE (Other); Centro Hospitalar de Leiria (Other); Centro Hospitalar do Oeste (Other); University of Coimbra (Other); IPM - Institute of Psychological Medicine, Faculty of Medicine, University of Coimbra (Unknown)
Responsible Party: Sponsor-Investigator, Julieta Azevedo, PhD student in Clinical Psychology, University of Coimbra
Organization: University of Coimbra (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BD/130116/2017_Pilot
Record Dates: First submitted 2021-03-07; First posted 2021-03-15 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder; DBT Skills; Recovery; Emotion Regulation
MeSH Terms: conditions — Bipolar Disorder; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: Participants are randomly distributed into 2 groups:
  Experimental Group: Treatment as Usual (Public health services and psychiatric support) + 1 Pre-session + 12 session DBT Skills Group Experimental Group Condition 2: Specialized support (Psychoeducation in Bipolar Disorder + Psychological support) + (1 Pre-session) 12 session DBT Skills group + TAU Control Group Condition 1: TAU + Waiting List
Who Masked: Outcomes Assessor
Masking Description: After the intervention participants will be interviewed by a health professional, not involved in the study, to assess feedback - regarding facilitators, program sessions, interest and usefulness.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): * Pre-treatment session + 12 Sessions Group Intervention
  * TAU - Treatment as usual (Psychiatric support through Public health system)
  Interventions: Behavioral: Dialectical Behavior Therapy - Skills
- Control Group (No Intervention): * TAU - Treatment as usual (Psychiatric support through Public health system)
  * Waiting list (will have access to the intervention program BI-REAL after the 3 month follow up assessment)

INTERVENTIONS:
Behavioral: Dialectical Behavior Therapy - Skills — Pre-treatment session + 12 sessions DBT Skills Group (only) intervention
  Other Names: Bi-REAL
  Arms: Experimental Group

SUMMARY:
Bipolar disorder (BD) is a serious mental disorder characterized by episodes of mania/hypomania and/or depression. Compared to the general population, these individuals present functional impairment, and life interference subclinical symptoms even between mood episodes, and higher mood instability and suicide rates with a lower quality of life. Given the chronic and phasic course of this disorder, patients are great consumers of health services and in Portugal there is no specialised psychotherapeutic approach to Bipolar Disorder, having pharmacological treatment alone as the main therapeutic response, and a considerable number of patients are not fully stabilized with drug treatments, experiencing residual symptoms. Although studies suggest that certain psychological therapies can be helpful for people experiencing full mood disorder episodes, or to reduce risk of future episodes, there are no gold standard and evidence-based psychological therapies for BD, and recent systematic reviews on psychosocial interventions for BD identify Dialectical-Behavior Therapy (DBT) as promising.

Our research is sustained in a recovery based perspective, which means we intend to develop a sense of hope, understanding, empowerment and work towards a meaningful and satisfying life, focusing on less clinical outcomes. Recovery is a concept that looks beyond the traditional clinical definitions which focus on reduced symptomatology, hospitalisation and medication compliance, and focuses on having a better sense of living even though you might have some clinical symptomatology.

DBT was developed as an approach for highly emotionally and behaviourally dysregulated people, and it has been referred as promising in BD patients. DBT aims to give individuals who experience quick and intense shifts in mood, skills to manage and regulate their emotions.

People with Bipolar Disorder can benefit from skills to regulate their emotions and interpersonal efficacy, which is frequently affected by mood changes, and therefore have a life worth living, feeling skillful and empowered to deal with challenges.

Our study aimed to develop a 12 session DBT-skills group adapting the sessions and skills to be used with this client group (Bi-REAL - Respond Effectively and Live mindfully).

This study aims to test acceptability, feasibility and efficacy of this 12 session DBT skills pilot randomized group intervention for patients with Bipolar Disorders.

DETAILED DESCRIPTION:
Bipolar disorder (BD) is a serious mental disorder characterized by episodes of mania or hypomania and depression, occurring with a typically cyclical course. In addition to mood instability, BD has been associated with significant functional impairment, lower quality of life, and higher rates of suicide compared to the general population. Prevalence of BD in Europe is of approximately 1%, with few evidences of gender differences. Despite the advances in pharmacological and non-pharmacological treatments, BD still entails multiple relapses. Prediction of the course and outcome continues to be challenging, and BD has been considered the sixth leading cause of disability-adjusted life years in the world, with high costs to society, patients and mental health services.

Even though the etiology of BD is still unclear, it is multifactorial with multiple genetic and environmental influences interacting with each other. Fewer studies have explored psychosocial factors in BD's development and maintenance, however, some risk factors have been identified, namely negative early experiences, family characteristics, and adverse life circumstances. Researchers also found significantly higher levels of childhood abuse and current internalized shame in BD individuals, when compared to a control group. It is also known that stressful life events possibly work as triggers in affective symptoms, and they are frequently stigmatized because of their condition, jeopardizing their social and work context.

Pharmacological interventions prevail as the primary management tool in BD, however, most patients are not fully stabilized on drug therapies alone and a large number of patients experience residual symptoms so that full functional recovery is uncommon. Hence, growing evidence and international guidelines support the need to use psychosocial interventions as adjuvant therapies to improve recovery in BD.

Our research is sustained in a recovery based perspective, which means we intend to develop a sense of hope, understanding, empowerment and work towards a meaningful and satisfying life, focusing on less clinical outcomes. Recovery is a concept that looks beyond the traditional clinical definitions which focus on reduced symptomatology, hospitalisation and medication compliance, and focuses on having a better sense of living even though you might have some clinical symptomatology.

The most empirically tested psychosocial interventions for BD include Psychoeducation (PE) and Cognitive-Behavioral Therapy (CBT) with supporting evidence of their efficacy. However, there are also contradictory findings, contesting the efficacy of CBT and PE, and that is why there is still no Goldstandard regarding BD psychosocial intervention. A recent review regarding empirically supported psychosocial interventions for BD, discusses promising findings regarding contextual therapies, namely Dialectical Behavior Therapy (DBT), and further research is encouraged.

DBT seems to be a promising approach to apply with BD, given its components for emotion regulation, and has already been found to reduce depressive and manic symptoms as well as to improve emotional dysregulation in BD groups. Based on the above-mentioned, further empirical research to clarify about contextual therapies efficacy (particularly DBT), for BD is essential and necessary which is why we constructed our 12-session skills intervention Bi-REAL (Respond Effectively and Live mindfully), based on some preliminary studies and suggested adaptations for DBT for Bipolar Disorder.

This study aims to test acceptability, feasibility and efficacy of this 12 session DBT skills pilot randomized group intervention for patients with Bipolar Disorders.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of bipolar disorder according to DSM-5 (BD-I, BD-II and Other (un)specified bipolar and related disorder) (APA, 2013), identified by psychiatrists or any assistant physician, and confirmed through CIBD;
* A history of two or more episodes of illness meeting DSM-5 criteria for mania, hypomania, major depressive disorder or mixed affective disorder, one of which must have been within 5 year of recruitment.
* Mood symptoms cause interference in their life (currently)
* Having a computer/tablet with access to internet, zoom installed, a microphone and camera.
* Living in Portugal and with good comprehension of Portuguese at a level sufficient to complete self-report instruments and clinical interview.

Exclusion Criteria:

* Active suicide ideation
* Bipolar disorder secondary to an organic cause;
* Continuous illicit substance misuse resulting in uncertain primary diagnosis;
* Acute episode of mania, hypomania or major depressive episode;
* Other high risk pervasive disorders such as Borderline Personality Disorder; persistent self-injury;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Sense of personal recovery | 6 months (from Baseline to 3-months follow-up)
  Assessed by the Bipolar Recovery Questionnaire (scores vary from 0-3600) higher scores mean a better outcome
Changes in quality of life | 6 months (from Baseline to 3-months follow-up)
  Assessed by Quality of Life Questionnaire for Bipolar Disorder (scores from 1-60) higher scores mean a better outcome

SECONDARY OUTCOMES:
Changes in activation and reactivity levels | 6 months (from Baseline to 3-months follow-up)
  Assessed through Multidimensional assessment of thymic states (0-200) continuum between Hypo-reactivity/Hyper-reactivity - median scores around 100 mean better outcome
Changes in Distress Tolerance | 6 months (from Baseline to 3-months follow-up)
  Assessed through Distress Tolerance Scale (1-75) - higher scores mean a better outcome
Changes in psychopathology symptoms | 6 months (from Baseline to 3-months follow-up)
  Assessed through Depression and Anxiety Stress Scale - lower scores mean a better outcome
Changes in Rumination | 6 months (from Baseline to 3-months follow-up)
  Assessed through Rumination-Reflexion Questionnaire (RRQ-10) lower scores mean a better outcome
Changes in symptoms interference with life | 6 months (from Baseline to 3-months follow-up)
  Assessed through semi-structured clinical interview for Bipolar Disorder (CIBD) lower scored mean less interference, thus better outcome

OTHER OUTCOMES:
Changes in Self-criticism | 6 months (from Baseline to 3-months follow-up)
  Assessed through Forms of self-criticizing/attacking and self-reassuring scale - lower scores in self-criticising mean a better outcome
Changes in Self-reassurance | 6 months (from Baseline to 3-months follow-up)
  Assessed through Forms of self-criticizing/attacking and self-reassuring scale - higher scores in self-reassurance mean a better outcome
Changes in Awareness and acceptance of experience | 6 months (from Baseline to 3-months follow-up)
  Assessed through Philadelphia Mindfulness Scale (PHLMS) - higher scores mean a better outcome
Changes in difficulties in emotional regulation | 6 months (from Baseline to 3-months follow-up)
  Assessed through Difficulties in Emotion Regulation Scale (DERS) - lower scores mean a better outcome
Changes in internal and external shame | 6 months (from Baseline to 3-months follow-up)
  Assessed through Internal and External Shame Scale (IESS) - lower scores mean a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Julieta M Azevedo, MS, Principal Investigator — University of Coimbra - CINEICC
Locations (1):
- Faculty of Psychology and Educational Sciences - University of Coimbra, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Azevedo, J., Macedo, A., Swales, M., & Castilho, P. (2019). A Dialectical Behaviour Therapy Skills' based intervention program for Bipolar Disorder - development of Bi-REAL. In proceedings 3ª Mostra de Doutoramento em Psicologia: - PsihDay 2019 (pp. 165-167). Coimbra; Psychologica. Accessible from https://doi.org/10.14195/1647-8606_63-1_9.
- [Background] DiRocco A, Liu L, Burrets M. Enhancing Dialectical Behavior Therapy for the Treatment of Bipolar Disorder. Psychiatr Q. 2020 Sep;91(3):629-654. doi: 10.1007/s11126-020-09709-6. PMID 32144641
- [Background] Balanza-Martinez V, Selva G, Martinez-Aran A, Prickaerts J, Salazar J, Gonzalez-Pinto A, Vieta E, Tabares-Seisdedos R. Neurocognition in bipolar disorders--a closer look at comorbidities and medications. Eur J Pharmacol. 2010 Jan 10;626(1):87-96. doi: 10.1016/j.ejphar.2009.10.018. Epub 2009 Oct 18. PMID 19836378
- [Background] Barnett JH, Smoller JW. The genetics of bipolar disorder. Neuroscience. 2009 Nov 24;164(1):331-43. doi: 10.1016/j.neuroscience.2009.03.080. Epub 2009 Apr 7. PMID 19358880
- [Background] Beynon S, Soares-Weiser K, Woolacott N, Duffy S, Geddes JR. Pharmacological interventions for the prevention of relapse in bipolar disorder: a systematic review of controlled trials. J Psychopharmacol. 2009 Jul;23(5):574-91. doi: 10.1177/0269881108093885. Epub 2008 Jul 17. PMID 18635701
- [Background] Cardoso Tde A, Farias Cde A, Mondin TC, da Silva Gdel G, Souza LD, da Silva RA, Pinheiro KT, do Amaral RG, Jansen K. Brief psychoeducation for bipolar disorder: impact on quality of life in young adults in a 6-month follow-up of a randomized controlled trial. Psychiatry Res. 2014 Dec 30;220(3):896-902. doi: 10.1016/j.psychres.2014.09.013. Epub 2014 Sep 28. PMID 25300245
- [Background] de Barros Pellegrinelli K, de O Costa LF, Silval KI, Dias VV, Roso MC, Bandeira M, Colom F, Moreno RA. Efficacy of psychoeducation on symptomatic and functional recovery in bipolar disorder. Acta Psychiatr Scand. 2013 Feb;127(2):153-8. doi: 10.1111/acps.12007. Epub 2012 Sep 4. PMID 22943487
- [Background] Dean BB, Gerner D, Gerner RH. A systematic review evaluating health-related quality of life, work impairment, and healthcare costs and utilization in bipolar disorder. Curr Med Res Opin. 2004;20(2):139-54. doi: 10.1185/030079903125002801. PMID 15006007
- [Background] Fowke A, Ross S, Ashcroft K. Childhood maltreatment and internalized shame in adults with a diagnosis of bipolar disorder. Clin Psychol Psychother. 2012 Sep;19(5):450-7. doi: 10.1002/cpp.752. Epub 2011 May 9. PMID 21557379
- [Background] Gama CS, Kunz M, Magalhaes PV, Kapczinski F. Staging and neuroprogression in bipolar disorder: a systematic review of the literature. Braz J Psychiatry. 2013 Mar;35(1):70-4. doi: 10.1016/j.rbp.2012.09.001. PMID 23567604
- [Background] Goldstein TR, Fersch-Podrat RK, Rivera M, Axelson DA, Merranko J, Yu H, Brent DA, Birmaher B. Dialectical behavior therapy for adolescents with bipolar disorder: results from a pilot randomized trial. J Child Adolesc Psychopharmacol. 2015 Mar;25(2):140-9. doi: 10.1089/cap.2013.0145. Epub 2014 Jul 10. PMID 25010702
- [Background] Van Dijk S, Jeffrey J, Katz MR. A randomized, controlled, pilot study of dialectical behavior therapy skills in a psychoeducational group for individuals with bipolar disorder. J Affect Disord. 2013 Mar 5;145(3):386-93. doi: 10.1016/j.jad.2012.05.054. Epub 2012 Aug 1. PMID 22858264
- [Background] Gomes BC, Abreu LN, Brietzke E, Caetano SC, Kleinman A, Nery FG, Lafer B. A randomized controlled trial of cognitive behavioral group therapy for bipolar disorder. Psychother Psychosom. 2011;80(3):144-50. doi: 10.1159/000320738. Epub 2011 Mar 3. PMID 21372622
- [Background] Goodwin GM, Haddad PM, Ferrier IN, Aronson JK, Barnes T, Cipriani A, Coghill DR, Fazel S, Geddes JR, Grunze H, Holmes EA, Howes O, Hudson S, Hunt N, Jones I, Macmillan IC, McAllister-Williams H, Miklowitz DR, Morriss R, Munafo M, Paton C, Saharkian BJ, Saunders K, Sinclair J, Taylor D, Vieta E, Young AH. Evidence-based guidelines for treating bipolar disorder: Revised third edition recommendations from the British Association for Psychopharmacology. J Psychopharmacol. 2016 Jun;30(6):495-553. doi: 10.1177/0269881116636545. Epub 2016 Mar 15. PMID 26979387
- [Background] Salcedo S, Gold AK, Sheikh S, Marcus PH, Nierenberg AA, Deckersbach T, Sylvia LG. Empirically supported psychosocial interventions for bipolar disorder: Current state of the research. J Affect Disord. 2016 Sep 1;201:203-14. doi: 10.1016/j.jad.2016.05.018. Epub 2016 May 14. PMID 27243619
- [Background] Linehan MM, Comtois KA, Murray AM, Brown MZ, Gallop RJ, Heard HL, Korslund KE, Tutek DA, Reynolds SK, Lindenboim N. Two-year randomized controlled trial and follow-up of dialectical behavior therapy vs therapy by experts for suicidal behaviors and borderline personality disorder. Arch Gen Psychiatry. 2006 Jul;63(7):757-66. doi: 10.1001/archpsyc.63.7.757. PMID 16818865
- [Background] Pini S, de Queiroz V, Pagnin D, Pezawas L, Angst J, Cassano GB, Wittchen HU. Prevalence and burden of bipolar disorders in European countries. Eur Neuropsychopharmacol. 2005 Aug;15(4):425-34. doi: 10.1016/j.euroneuro.2005.04.011. PMID 15935623
- [Background] Todd NJ, Jones SH, Lobban FA. "Recovery" in bipolar disorder: how can service users be supported through a self-management intervention? A qualitative focus group study. J Ment Health. 2012 Apr;21(2):114-26. doi: 10.3109/09638237.2011.621471. Epub 2011 Dec 5. PMID 22142324
- [Background] Morrison AP, Law H, Barrowclough C, Bentall RP, Haddock G, Jones SH, Kilbride M, Pitt E, Shryane N, Tarrier N, Welford M, Dunn G. Psychological approaches to understanding and promoting recovery in psychosis and bipolar disorder: a mixed-methods approach. Southampton (UK): NIHR Journals Library; 2016 May. Available from http://www.ncbi.nlm.nih.gov/books/NBK361044/ PMID 27170958
- [Background] Wright K, Dodd A, Warren FC, Medina-Lara A, Taylor R, Jones S, Owens C, Javaid M, Dunn B, Harvey JE, Newbold A, Lynch T. The clinical and cost effectiveness of adapted dialectical behaviour therapy (DBT) for bipolar mood instability in primary care (ThrIVe-B programme): a feasibility study. Trials. 2018 Oct 16;19(1):560. doi: 10.1186/s13063-018-2926-7. PMID 30326960
- [Background] Jones S, Mulligan LD, Higginson S, Dunn G, Morrison AP. The bipolar recovery questionnaire: psychometric properties of a quantitative measure of recovery experiences in bipolar disorder. J Affect Disord. 2013 May;147(1-3):34-43. doi: 10.1016/j.jad.2012.10.003. Epub 2012 Nov 22. PMID 23182591

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-31): https://cdn.clinicaltrials.gov/large-docs/51/NCT04797351/Prot_SAP_000.pdf